CLINICAL TRIAL: NCT01485679
Title: Evaluation of 18 Fluoro-deoxy-glucose Positrons Emission Tomography Combined With Computed Tomography (18-FDG TEP-CT ) in the Diagnosis of the Degeneration of Intraductal Papillary Mucinous Tumor of the Pancreas
Brief Title: 18 Fluoro-deoxy-glucose Positrons Emission Tomography Combined With Computed Tomography (18-FDG TEP-CT ) in the Diagnosis of the Degeneration of Intraductal Papillary Mucinous Tumor of the Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD/10/06-P
Record Dates: First submitted 2011-08-26; First posted 2011-12-05 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2015-10

CONDITIONS: Tumor
Keywords: 18 fluoro deoxy glucose positrons emission tomography combined with computed tomography,; Patients with intraductal papillary mucinous tumor of the pancreas; intraductal papillary mucinous; pancreas
MeSH Terms: conditions — Neoplasms

ARMS (1):
- positrons emission tomography (Experimental)
  Interventions: Other: 18 fluoro-deoxy-glucose positrons emission tomography combined with computed tomography

INTERVENTIONS:
Other: 18 fluoro-deoxy-glucose positrons emission tomography combined with computed tomography — 18 fluoro-deoxy-glucose positrons emission tomography combined with computed tomography

SUMMARY:
The aim of the study is to evaluate whether the TEP-CT can be sensitive and specific in identifying degenerated intraductal papillary mucinous tumor of the pancreas.The results will be compared to those obtained by the pathological analysis of the removed piece of pancreas.

DETAILED DESCRIPTION:
Before surgery is undertaken, a 18 fluoro-deoxy-glucose positrons emission tomography combined with computed tomography (18-FDG TEP-CT ) will be performed. The primary outcome of this study is to compare results of the TEP-CT with those obtained by the pathological analysis of the removed piece of pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age equal or above 18
* Patients diagnosed with intraductal papillary mucinous tumor with surgical indication and for whom it will be possible to have the pathological analysis of the removed piece of pancreas.
* if woman being of childbearing potential, woman taking contraceptive measures
* Patient able to understand benefits and risks of protocol
* Subject affiliated to French health insurance (Social Security)
* Informed consent form signed

Exclusion Criteria:

* Patients not fulfilling inclusion criteria
* Pancreatic surgery or radiotherapy in the pancreatic zone within 4 the months preceding the TEP-CT
* Chemotherapy within 2 the months preceding the TEP-CT
* Acute pancreatitis within 2 the months preceding the TEP-CT
* Pregnant women or breast-feeding women refusing to temporary stop it
* Diabetes not equilibrated (checked by glycemia and glycosylated hemoglobin (HbA1c) at inclusion) or Fasting blood glucose below 7mmol/L (126 g/L before the TEP)
* Patients with claustrophobia
* Patients not accepted under the anesthesia point of view

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Specificity of TEP-CT to point out malignant lesions in pancreas, the gold standard being the anatomopathological analysis of the piece of pancreas removed during the surgery. | 3 months
  TEP-CT of the different 5 parts of the pancreas (head, uncus, isthmi, body and tail) will be interpreted by nuclearity Doctors. TEP-CT will be considered positive if there is a pathological fixation of the 18-FDG , defined as any focal or diffuse fixation of 18-FDG above the background level of fixation in the pancreas.
  The anatomopathological analysis of the piece of pancreas removed during the ablative surgery will be considered as positive if the degree of dysplasia seen for each part of the pancreas is "infiltrating carcinoma".
  Results will then be compared in term of specificity.

SECONDARY OUTCOMES:
Sensitivity of TEP-CT to point out malignant lesions in pancreas, the gold standard being the anatomopathological analysis of the piece of pancreas removed during the surgery. | 3 months
  TEP-CT of the different 5 parts of the pancreas (head, uncus, isthmi, body and tail) will be interpreted by nuclearity Doctors. TEP-CT will be considered positive if there is a pathological fixation of the 18-FDG , defined as any focal or diffuse fixation of 18-FDG above the background level of fixation in the pancreas.
  The anatomopathological analysis of the piece of pancreas removed during the ablative surgery will be considered as positive if the degree of dysplasia seen for each part of the pancreas is "infiltrating carcinoma".
  Results will then be compared in term of sensitivity.
Comparison of specificity of the TEP-CT to detect malignant lesions in pancreas versus specificity of conventional devices, the gold standard being the anatomopathological analysis results | 3 months
  Result of conventional devices (such as computed tomography, magnetic resonance cholangiopancreatography or endoscopic ultrasound) will be considered positive if diagnosis is "malignant lesion" or "probable malignant lesion". The 5 parts of the pancreas will be examined.
Number of patients for which metastasis will be detected through TEP-CT and confirmed by biopsy and/or conventional specific device | 3 months

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU Nord, Amiens, France
  - Maison de Haut Lévêque CHU, Bordeaux, France
  - Hôpital Beaujon APHP, Clichy, France
  - Hôpital C Huriez, Lille, France
  - Hospices Civils de Lyon, Lyon, France
  - Institut Paoli Calmettes, Marseille, France
  - CHU Nord, Marseille, France
  - CHU, Nantes, France
  - CHU Hôpital Pontchaillou, Rennes, France
  - Hôpital de Hautepierre, Strasbourg, France
  - Hôpital St-Antoine, Paris
  - CHU Rangueil, Toulouse